CLINICAL TRIAL: NCT03329729
Title: Non-interventional, Multicenter Clinical Trial to Investigate the Efficacy of Rosuvastatin in Patients With Hyperlipidemia and Other Cardiovascular Risk Factors.
Brief Title: PLATOREL® STUDY IN CARDIOVASCULAR RISΚ ASSESMENT
Acronym: PLATINUM
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-RSV-EL-78
Record Dates: First submitted 2017-10-24; First posted 2017-11-06 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2018-12

CONDITIONS: Dyslipidemias; Hyperlipidemias; Risk Factor, Cardiovascular; Quality of Life
MeSH Terms: conditions — Dyslipidemias; Hyperlipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyperlipidemic patients
  Interventions: Other: Rosuvastatin

INTERVENTIONS:
Other: Rosuvastatin — Hyperlipidemic patients treated with rosuvastatin

SUMMARY:
Dyslipidemias are a major risk factor for the onset of cardiovascular disease, while early diagnosis and appropriate treatment approaches significantly reduce cardiovascular morbidity and mortality.

The aim is to provide revised Greek guidelines for the diagnosis and treatment of dyslipidaemias.

The lipids of the human body are cholesterol (it is used to synthesize cell membranes, adrenal hormones and gonads and is a component of bile) and triglycerides (used as a fuel and as a storage of energy in adipose tissue). Dyslipidemias are disorders (quantitative or qualitative) of the metabolism of lipoprotein particles [low density lipoproteins (LDL), chylomic, high density lipoproteins (HDL), very low density lipoproteins (VLDL)] that carry lipids into the body.

Primary prevention in subjects aged 40-65 years with no known clinical atherosclerotic disease and without diabetes or chronic renal disease should evaluate the likelihood of a fatal cardiovascular event over the next 10 years. For this purpose, it is recommended to use the Greek version of the SCORE of the Hellenic Heart SCORE.

DETAILED DESCRIPTION:
Rosuvastatin is a selective and competitive inhibitor of 3-hydroxy-3-methylglutaric coenzyme A (HMG-CoA), an enzyme regulating the rate of cholesterol synthesis. Its main area of action is the liver.

* In cases of primary hypercholesterolaemia (type IIa, including familial hypercholesterolemia heterozygote) or mixed dyslipidaemia (type IIb) as a supplement to diet when dietary and other non-medication responses are inadequate.
* In cases of homozygous familial hypercholesterolemia (HoFH), as a supplement to the diet and other lipid-lowering treatments.
* In cases of slowing the progression of atherosclerosis. It is indicated as a supplemental treatment of the diet in lowering the total cholesterol (Total C) and LDL-C values.
* In patients with hypertriglyceridaemia (excess triglycerides in the blood). Dosage and route of administration
* In hyperlipidemia, mixed dyslipidaemia, hypertriglyceridaemia, and slowing the progression of atherosclerosis, the recommended starting dose is 10 mg once a day.
* In homozygous familial hypercholesterolemia, the recommended starting dose is 20 mg once a day.
* In Asian patients, the recommended starting dose is 5mg once a day.
* In patients receiving ciclosporin, the dose of rosuvastatin should be set at 5 mg, while those taking the combination of Lopinavir

ELIGIBILITY:
Inclusion Criteria:

* Outpatient Patients who are monitored at an external hospital for lipids, hypercholesterolemia, diabetes,
* Male or female
* Eligible ages for study: 18 - 99 years
* Patients diagnosed with hypercholesterolemia who are to receive Rosuvastatin according to established clinical practice
* Acquired cardiovascular disease from invasive or non-invasive examinations (such as coronary angiography, nuclear medicine, stress echocardiography, carotid plaque ultrasound), previous myocardial infarction, ACS, coronary revascularization (PCI, CABG), and other arterial revascularization, ischemic cerebrovascular accident, peripheral arterial disease (PAD) Diabetes mellitus (type 1 or type 2) with one or more cardiovascular risk factors orand target organ damage (such as microalbuminuria: 30-300 mg Patients already diagnosed with hypercholesterolemia and non-regulated who are going to receive Rosuvastatin according to established clinical practice
* Patients who have fully understood the study protocol and have signed the consent document
* Compliance with study procedures

Exclusion Criteria:

* Patients <18 years
* Hypersensitivity to Rosuvastatin or to any of the excipients
* Women in gestation or lactation
* Patients who have not fully understood the study protocol and have not signed the consent document

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dyslipidemia and other risk factors treated with rosuvastatin
Sampling Method: Non-Probability Sample
Enrollment: 4700 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Time to achieve LDL-C goal | 6 months
  To evaluate the efficacy of rosuvastatin in patients with hypercholesterolemia in achieving the target lipid level (LDL-C, HDL-C, T-CHOL) in patients' blood plasma

SECONDARY OUTCOMES:
CV Risk Factor | 6 months
  Assessing the Cardiovascular Disease Index - 10-year cardiovascular risk
Quality of Life | 6 months
  Assessing Quality of Life in patients with hypercholesterolemia and other risk factors by EQ-5D questionnaire. The EQ- 5D is a descriptive, generic instrument that has also been validated for the Greek population and consists of two parts.25 The first part is a descriptive system of five dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The second part consists of a visual analogue scale (VAS), the EQ-VAS, that asks respondents to self-rate themselves on a thermometer-like grading system in order to capture variations in health states. EQ-5D health state valuations may be converted into a single summary index by applying an algorithm that attaches values to each of the levels in each dimension. Value sets have been derived for the EQ-5D scores in several countries using either the VAS or the time trade-off (TTO) valuation technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Agia Olga Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Catapano AL, Graham I, De Backer G, Wiklund O, Chapman MJ, Drexel H, Hoes AW, Jennings CS, Landmesser U, Pedersen TR, Reiner Z, Riccardi G, Taskinen MR, Tokgozoglu L, Verschuren WMM, Vlachopoulos C, Wood DA, Zamorano JL, Cooney MT; ESC Scientific Document Group. 2016 ESC/EAS Guidelines for the Management of Dyslipidaemias. Eur Heart J. 2016 Oct 14;37(39):2999-3058. doi: 10.1093/eurheartj/ehw272. Epub 2016 Aug 27. No abstract available. PMID 27567407
- [Background] European Association for Cardiovascular Prevention & Rehabilitation; Reiner Z, Catapano AL, De Backer G, Graham I, Taskinen MR, Wiklund O, Agewall S, Alegria E, Chapman MJ, Durrington P, Erdine S, Halcox J, Hobbs R, Kjekshus J, Filardi PP, Riccardi G, Storey RF, Wood D; ESC Committee for Practice Guidelines (CPG) 2008-2010 and 2010-2012 Committees. ESC/EAS Guidelines for the management of dyslipidaemias: the Task Force for the management of dyslipidaemias of the European Society of Cardiology (ESC) and the European Atherosclerosis Society (EAS). Eur Heart J. 2011 Jul;32(14):1769-818. doi: 10.1093/eurheartj/ehr158. Epub 2011 Jun 28. PMID 21712404
- [Background] Authors/Task Force Members:; Catapano AL, Graham I, De Backer G, Wiklund O, Chapman MJ, Drexel H, Hoes AW, Jennings CS, Landmesser U, Pedersen TR, Reiner Z, Riccardi G, Taskinen MR, Tokgozoglu L, Verschuren WM, Vlachopoulos C, Wood DA, Zamorano JL. 2016 ESC/EAS Guidelines for the Management of Dyslipidaemias: The Task Force for the Management of Dyslipidaemias of the European Society of Cardiology (ESC) and European Atherosclerosis Society (EAS) Developed with the special contribution of the European Assocciation for Cardiovascular Prevention & Rehabilitation (EACPR). Atherosclerosis. 2016 Oct;253:281-344. doi: 10.1016/j.atherosclerosis.2016.08.018. Epub 2016 Sep 1. No abstract available. PMID 27594540
- [Background] Task Force for the management of dyslipidaemias of the European Society of Cardiology (ESC) and the European Atherosclerosis Society (EAS); Catapano AL, Reiner Z, De Backer G, Graham I, Taskinen MR, Wiklund O, Agewall S, Alegria E, Chapman MJ, Durrington P, Erdine S, Halcox J, Hobbs R, Kjekshus J, Perrone Filardi P, Riccardi G, Storey RF, Wood D; ESC Committee for Practice Guidelines 2008-2010 and 2010-2012 Committees. ESC/EAS Guidelines for the management of dyslipidaemias: the Task Force for the management of dyslipidaemias of the European Society of Cardiology (ESC) and the European Atherosclerosis Society (EAS). Atherosclerosis. 2011 Jul;217 Suppl 1:S1-44. doi: 10.1016/j.atherosclerosis.2011.06.012. No abstract available. PMID 21723445
- [Background] Hamm CW, Bassand JP, Agewall S, Bax J, Boersma E, Bueno H, Caso P, Dudek D, Gielen S, Huber K, Ohman M, Petrie MC, Sonntag F, Uva MS, Storey RF, Wijns W, Zahger D; ESC Committee for Practice Guidelines. ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: The Task Force for the management of acute coronary syndromes (ACS) in patients presenting without persistent ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2011 Dec;32(23):2999-3054. doi: 10.1093/eurheartj/ehr236. Epub 2011 Aug 26. No abstract available. PMID 21873419
- [Background] Panagiotakos DB, Fitzgerald AP, Pitsavos C, Pipilis A, Graham I, Stefanadis C. Statistical modelling of 10-year fatal cardiovascular disease risk in Greece: the HellenicSCORE (a calibration of the ESC SCORE project). Hellenic J Cardiol. 2007 Mar-Apr;48(2):55-63. PMID 17489342
- [Background] Panagiotakos DB, Georgousopoulou EN, Fitzgerald AP, Pitsavos C, Stefanadis C. Validation of the HellenicSCORE (a Calibration of the ESC SCORE Project) Regarding 10-Year Risk of Fatal Cardiovascular Disease in Greece. Hellenic J Cardiol. 2015 Jul-Aug;56(4):302-8. PMID 26233769
- [Background] Pitsavos C, Panagiotakos DB, Chrysohoou C, Stefanadis C. Epidemiology of cardiovascular risk factors in Greece: aims, design and baseline characteristics of the ATTICA study. BMC Public Health. 2003 Oct 20;3:32. doi: 10.1186/1471-2458-3-32. PMID 14567760
- [Background] Panagiotakos DB, Pitsavos C, Manios Y, Polychronopoulos E, Chrysohoou CA, Stefanadis C. Socio-economic status in relation to risk factors associated with cardiovascular disease, in healthy individuals from the ATTICA study. Eur J Cardiovasc Prev Rehabil. 2005 Feb;12(1):68-74. PMID 15703509
- [Background] Kontodimopoulos N, Pappa E, Niakas D, Tountas Y. Validity of SF-12 summary scores in a Greek general population. Health Qual Life Outcomes. 2007 Sep 28;5:55. doi: 10.1186/1477-7525-5-55. PMID 17900374